CLINICAL TRIAL: NCT06921772
Title: The Effects of Proprioceptive Neuromuscular Facilitation Stretching Exercises on Anaerobic Power and Motor Performance in Adolescent Male Volleyball Players: A Randomized Controlled Trial
Brief Title: The Effects of PNF Stretching on Anaerobic Power and Motor Performance in Adolescent Male Volleyball Players
Acronym: PNF-VMVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zarife Pancar (Other)
Responsible Party: Sponsor-Investigator, Zarife Pancar, Associate Professor, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GAUN-SBF-PANCAR-05
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Motor Performance; Anaerobic Power; Flexibility; Stretching
Keywords: Volleyball; Adolescent Athletes; PNF Stretching; Exercise Intervention
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: The study used a parallel assignment model with two arms. Participants were randomly assigned to either the experimental group, which received PNF stretching exercises in addition to regular training, or the control group, which continued only with standard volleyball training.
Who Masked: Outcomes Assessor
Masking Description: The assessor responsible for outcome measurements was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PNF Stretching Group (Experimental): Participants in this group performed proprioceptive neuromuscular facilitation (PNF) stretching exercises three times per week for six weeks, in addition to their regular volleyball training.
  Interventions: Behavioral: PNF Stretching Exercise
- Control Group (No Intervention): Participants in this group continued with their regular volleyball training without any additional intervention.

INTERVENTIONS:
Behavioral: PNF Stretching Exercise — Proprioceptive Neuromuscular Facilitation (PNF) stretching exercises were applied three times per week for six weeks. The intervention included contract-relax and hold-relax techniques targeting lower extremity muscle groups, conducted in addition to regular volleyball training.
  Arms: PNF Stretching Group

SUMMARY:
This randomized controlled study aimed to examine the effects of proprioceptive neuromuscular facilitation (PNF) stretching exercises on anaerobic power and motor performance in adolescent male volleyball players. Eighteen participants aged 15 to 17 years were randomly assigned to an experimental group and a control group. The experimental group performed PNF stretching exercises three times per week for six weeks, in addition to their regular volleyball training. The control group continued their standard volleyball training without PNF stretching. Outcome measures included anaerobic power, flexibility, balance, speed, push-up, and crunch tests. The study hypothesizes that PNF stretching will improve motor performance indicators in adolescent athletes.

DETAILED DESCRIPTION:
This clinical trial investigates the effects of a six-week proprioceptive neuromuscular facilitation (PNF) stretching intervention on motor performance in adolescent male volleyball players. A total of 18 participants with at least 6 months of volleyball training experience were randomly divided into two groups: the experimental group (n=9) and the control group (n=9). The experimental group received PNF stretching exercises in addition to their routine training three times per week for six weeks, while the control group continued only with their routine training.

The main outcome measures were anaerobic power (Margaria-Kalamen Test), flexibility (Sit-and-Reach Test), balance (Flamingo Balance Test), speed (20 m sprint), upper body strength (Push-up Test), and core strength (Crunch Test). Pre- and post-test evaluations were conducted. This study contributes to the growing body of literature on flexibility and functional performance development in adolescent athletes and aims to support evidence-based training practices in sports sciences.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Aged between 15 and 17 years
* At least 2 years of volleyball training experience
* Voluntarily agreeing to participate in the study
* No recent musculoskeletal injuries (in the last 6 months)

Exclusion Criteria:

* Participants with any diagnosed neurological or cardiovascular disorder
* Current use of performance-enhancing drugs or supplements
* History of lower extremity surgery
* Inability to complete the training or testing sessions
* Failure to provide written informed consent

Ages: 15 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only biologically male participants are eligible to participate in this study.
Enrollment: 18 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Anaerobic Power (Margaria-Kalamen Test) | Baseline and after 6-week intervention
  Anaerobic power will be evaluated using the Margaria-Kalamen test, which measures power output based on the time taken to run up a staircase. The test will be conducted at baseline and after 6 weeks.
Hamstring Flexibility (Sit-and-Reach Test) | Baseline and after 6-week intervention
  Hamstring flexibility will be measured with the Sit-and-Reach test. Participants sit on the floor with legs extended and reach forward. The distance reached is recorded in centimeters.
Static Balance Performance | Baseline and after 6-week intervention
  Static balance will be measured by having participants stand on one leg for a defined duration without support. Performance will be evaluated based on duration of balance and postural stability.
Sprint Performance (20-m Sprint Test) | Baseline and after 6-week intervention
  Speed performance will be measured using the 20-meter sprint test. Participants will run 20 meters at maximal effort, and the time taken will be recorded in seconds.
Upper Body Endurance (Push-Up Test) | Baseline and after 6-week intervention
  Upper body muscular endurance will be evaluated by counting the number of push-ups performed within 30 seconds.
Core Endurance (Crunch Test) | Baseline and after 6-week intervention
  Core endurance will be assessed by counting the number of crunches a participant can perform in 30 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Faculty of Sport Sciences, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared in an anonymized format. No personally identifiable information will be included. Data will be limited to outcome measures and relevant variables necessary for reproducibility and secondary analyses by qualified researchers upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available beginning 6 months after publication of the results and will be available for 5 years.